CLINICAL TRIAL: NCT06492070
Title: Prevention of Paclitaxel-Induced Peripheral Neuropathy: Randomized Trial of Cryocompression With or Without Cilostazol
Brief Title: Cryocompression With or Without Cilostazol for the Prevention of Paclitaxel-induced Neuropathy in Patients With Gynecological Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Modesitt, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007242; NCI-2024-03905 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007242 (Other: Emory University Hospital/Winship Cancer Institute); Winship6141-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cervical Carcinoma; Fallopian Tube Carcinoma; Malignant Solid Neoplasm; Malignant Uterine Neoplasm; Ovarian Carcinoma; Primary Peritoneal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Vulvar Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Cilostazol; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 2 (cryocompression) (Experimental): Patients receive paclitaxel infusions QD and receive cryocompression therapy with cooling compression wraps TID for 15 minutes before, during, and after receiving paclitaxel infusions on day 1 of each cycle. Treatment with paclitaxel continues up to 6-9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Cryocompression Therapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm A (cryocompression and cilostazol) (Experimental): Patients receive paclitaxel infusion QD and receive cryocompression therapy with cooling compression wraps TID over 15 minutes before, during, and after receiving paclitaxel infusion on day 1 of each cycle. Patients also receive cilostazol PO BID beginning with their first paclitaxel infusion continuing until 2 weeks after the final paclitaxel infusion. Treatment with paclitaxel continues for up to 6-9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cilostazol; Device: Cryocompression Therapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm C (standard of care) (Active Comparator): Patients undergo standard of care throughout the study.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm C (standard of care)
Drug: Cilostazol — Given PO
  Other Names: Pletal
  Arms: Arm A (cryocompression and cilostazol)
Device: Cryocompression Therapy — Undergo cryocompression therapy
  Arms: Arm 2 (cryocompression); Arm A (cryocompression and cilostazol)
Drug: Paclitaxel — Given by infusion
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm 2 (cryocompression); Arm A (cryocompression and cilostazol)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
The phase II trial evaluates the effectiveness of cryocompression therapy alone or in combination with cilostazol in preventing paclitaxel-induced peripheral neuropathy (numbness, pain or tingling in the feet and hands) for patients with gynecologic cancers. Peripheral neuropathy is a common side effect of many chemotherapeutic agents, including paclitaxel. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Cryocompression is a therapy that combines compression garments or dressings with cooling of the treated area. Cilostazol is in a class of medications called platelet-aggregation inhibitors (antiplatelet medications). It works by improving blood flow to the legs. Giving cilostazol together with cryocompression may be safe and tolerable in treating patients with gynecological cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantify the incidence and severity of peripheral neuropathy in women treated with paclitaxel for gynecologic malignancies in conjunction with cryocompression and to assess the impact of cilostazol on the development of peripheral neuropathy. (ARM A and ARM B) II. To quantify the baseline post-chemotherapy neuropathy rates among patients with gynecologic malignancies following standard clinical care practices according to their treating physician. (ARM C)

SECONDARY OBJECTIVES:

I. To estimate the potential impact of cilostazol on quality of life related to chemotherapy-induced peripheral neuropathy.

II. To estimate the potential impact of cilostazol on the need for pharmacologic symptom management for peripheral neuropathy.

III. To estimate the potential impact of cilostazol on chemotherapy dose reductions and delays due to peripheral neuropathy.

IV. To assess the safety of using cilostazol in conjunction with chemotherapy regimens with platinum/paclitaxel with or without VEGF inhibition, with or without immunotherapy, and with or without HER2-directed therapy.

OUTLINE: Participants are assigned to 1 of 3 arms.

ARM A: Patients receive paclitaxel infusion once daily (QD) and receive cryocompression therapy with cooling compression wraps three times daily (TID) over 15 minutes before, during, and after receiving paclitaxel infusion on day 1 of each cycle. Patients also receive cilostazol orally (PO) twice daily (BID) beginning with their first paclitaxel infusion continuing until 2 weeks after the final paclitaxel infusion. Treatment with paclitaxel continues for up to 6-9 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive paclitaxel infusions QD and receive cryocompression therapy with cooling compression wraps TID for 15 minutes before, during, and after receiving paclitaxel infusions on day 1 of each cycle. Treatment with paclitaxel continues for up to 6-9 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Patients undergo standard of care throughout the study.

After completion of study treatment, patients are followed up at 30 days and then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR ARMS A and B:
* Age 18 years or older
* Diagnosis of uterine, ovarian/fallopian tube/primary peritoneal, cervical, or vulvar cancer and planned chemotherapy regimen of 6-9 cycles of paclitaxel and carboplatin or cisplatin with or without VEGF inhibition, with or without immunotherapy, and with or without HER2-directed therapy
* Eastern Cooperative Oncology Group performance status from 0 to 2
* ARM C: Age 18 years or older
* ARM C: Diagnosis of uterine, ovarian/fallopian tube/primary peritoneal, cervical, or vulvar cancer and completion of 6-9 cycles of a chemotherapy regimen consisting of paclitaxel and carboplatin or cisplatin with or without VEGF inhibition, with or without immunotherapy, and with or without HER2-directed therapy within the last 3 months
* ARM C: Eastern Cooperative Oncology Group performance status from 0 to 2

Exclusion Criteria:

* EXCLUSION CRITERIA FOR ARMS A and B:
* Any patient unable and/or unwilling to cooperate with all study protocols
* Previous treatment with paclitaxel
* Patients with baseline pre-chemotherapy neuropathy requiring pharmacologic treatment
* Diabetes mellitus with hemoglobin A1c >7.0
* Hepatic impairment, moderate to severe (Class B & C by Child-Pugh score)

  * Slight or moderate malignant ascites alone will not be considered indicative of hepatic impairment in the absence of other evidence of hepatic disease
* Raynaud's phenomenon
* Active wounds on the hands or feet
* High risk uncontrolled arrhythmias
* Ischemic heart disease
* Inadequate bone marrow function with white blood count < 4,000/mm^3 and platelet count < 100,000/mm^3
* Inadequate liver function with serum total bilirubin >= 1.5mg/dL
* Inadequate renal function with serum creatinine >= 1.5mg/dL
* On one or more antiplatelet therapies excluding acetylsalicylic acid
* Hypersensitivity (e.g. anaphylaxis, angioedema) to cilostazol or any components of cilostazol
* Pregnant and nursing patients

  * Patients enrolled in this study who have the potential to become pregnant (have an intact uterus, ovary(ies), and fallopian tube(s), have not entered menopause, and have regular menses) are required to utilize reliable contraception such as celibacy, hormonal contraception (oral pills, implant, injection, ring or patch), intrauterine device (IUD), condom and/or diaphragm with spermicide
* Incarcerated patients
* Patients unable to consent for themselves, due to cognitive impairment or other reason
* Patients with contraindications to cilostazol
* Any patient who does not meet criteria to receive chemotherapy
* ARM C: Any patient unable and/or unwilling to cooperate with all study protocols
* ARM C: Previous treatment with paclitaxel
* ARM C: Patients with baseline pre-chemotherapy neuropathy requiring pharmacologic treatment
* ARM C: Diabetes mellitus with hemoglobin A1c >7.0
* ARM C: Pregnant patients
* ARM C: Incarcerated patients
* ARM C: Patients unable to consent for themselves, due to cognitive impairment or other reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in sensation and vibration objective neuropathy scores (Arms A and B) | At 1 month post chemotherapy completion and at 6 months and 12 months
  Specifically, the primary outcome will be the proportion of patients with abnormal vibration sensation times on at least one great toe or index finger assessed by a validated Neuropathy Assessment instrument. Will be compared between treatment groups (Arms A and B) using a chi-square test of independence.
Rates of impaired sensation and vibration on objective neuropathy testing and ≥ Grade 2 neuropathy among patients who recently completed paclitaxel treatment with standard of care treatment protocols (Arm C) | At 1 month post chemotherapy completion and at 6 months and 12 months
  The proportion of patients in Arm C will be tabulated with associated Clopper-Pearson 95% confidence intervals.

SECONDARY OUTCOMES:
Difference in sensation and vibration objective neuropathy scores | At 1 month post chemotherapy completion and at 6 months and 12 months
  Specifically, the outcome of interest will be the proportion of patients with abnormal vibration sensation times on at least one great toe or index finger assessed by a validated Neuropathy Assessment instrument. Will be compared between treatment groups using a chi-square test of independence.
Difference in >= grade 2 neuropathy between the two study arms | At 1 month post chemotherapy completion and at 6 months and 12 months
  Will be compared between treatment groups using a chi-square test of independence.
Changes in Functional Assessment of Cancer Therapy/Gynecologic Oncology Group- Neurotoxicity (FACT/GOG-NTX) scores | At 1 month post chemotherapy completion and at 6 months and 12 months
  Will be compared between treatment groups using a chi-square test of independence, as will the proportion of patients experiencing a clinically significant change in FACT/GOG-O-NTX neuropathy scores. Proportion of patients with a clinically significant change in scores (change of 10% or more from baseline) will also be determined.
Differences in the rate of patients starting new pharmacologic therapy for peripheral neuropathy while receiving paclitaxel chemotherapy | At 1 month post chemotherapy completion and at 6 months and 12 months
Differences in the rate of patients requiring paclitaxel dose reductions or chemotherapy delays due to peripheral neuropathy | At 1 month post chemotherapy completion and at 6 months and 12 months
Rate of grade 3 adverse events | At 1 month post chemotherapy completion and at 6 months and 12 months
  Will be tabulated by group according to Common Terminology Criteria for Adverse Events Grade, System Organ Class and relation to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan C Modesitt, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia